CLINICAL TRIAL: NCT05491668
Title: Physiological Assessment of Severe Coronary Stenosis for Informing Planned PCI (REFINE PCI)
Brief Title: Physiological Assessment of Severe Coronary Stenosis for Informing Planned PCI
Acronym: REFINE PCI
Status: Recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Opsens, Inc. (Industry)
Responsible Party: Principal Investigator, Eric A Osborn, MD, PhD, Director, Interventional Cardiology Fellowship, Beth Israel Deaconess Medical Center; Assistant Professor of Medicine, Harvard Medical School, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000479
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Invasive physiology; Angiography; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Coronary Physiology Assessment: Patients undergoing coronary angiogram who are found to have >/= 70% coronary stenosis and planned for percutaneous coronary intervention (PCI)/stent placement, will undergo pre and post PCI invasive physiologic assessment with a coronary pressure-sensing wire (OpSens OptoWire III) using non-hyperemic pressure ratio (NHPR) indices (diastolic pressure ratio [dPR]). Both the patient and interventional cardiologist will be blinded to the results of the invasive physiologic assessment. Angiogram co-registration will be performed on pullback of coronary pressure-sensing wire.
  Interventions: Diagnostic Test: Non-hyperemic pressure ratio assessment pre and post PCI

INTERVENTIONS:
Diagnostic Test: Non-hyperemic pressure ratio assessment pre and post PCI — Pre and post PCI invasive physiologic assessment
  Other Names: OpSens OptoWire III

SUMMARY:
Traditionally, the severity of a blockage (stenosis) in a coronary artery has been determined by visual angiographic assessment of the diameter of the artery at the level of a blockage compared to a normal healthy area of the same artery. With the advent of invasive physiological testing to assess coronary blood flow, multiple clinical trials have demonstrated a clinical benefit to a physiology-guided percutaneous coronary intervention (PCI) approach. However, despite this and the potential for significant variation in the interpretation of coronary artery stenosis severity by visual angiography alone to guide PCI, invasive physiologic indices remain significantly under-utilized.

The purpose of this study is to investigate the physiologic significance of coronary lesions deemed angiographically severe by visual estimation that are planned for PCI. The investigators plan to perform blinded physiologic assessment pre and post PCI. The primary aim of the study is to determine whether a subset of lesions visually estimated as severe by angiography treated with stent placement/PCI may in fact not be physiologically significant when assessed invasively, and thus PCI could safely be deferred in these patients. A secondary aim is to evaluate physiologic assessment post PCI to detect residual ischemia that could be utilized to optimize stent placement.

DETAILED DESCRIPTION:
Invasive physiological assessment via both resting and hyperemic indices has been shown to correlate with clinical outcomes in multiple controlled clinical trials. The traditional approach for the use of physiologic assessment has been in the context of angiographic intermediate lesions, defined as a stenosis between 40-70% stenosis by visual assessment, however it is plausible it could also be used in the context of coronary artery stenosis deemed severe (>70%) by visual assessment given the clear limitations to an angiography approach alone. A subgroup analysis of the Fractional Flow Reserve Versus Angiography in Multivessel Evaluation (FAME trial) suggested that only 80% of the lesions deemed significant (70-90% diameter stenosis) by angiography were also flow limiting by invasive physiology. Recent studies have further revealed that the role of physiologic assessments can be expanded to optimize the results after PCI by detecting residual ischemia both in the form of diffuse and focal lesions.

With advances in technology in recent years, the current generation of coronary pressure-sensing wires now exhibit performances similar to that of traditional work-horse wires. This, coupled with the advent of non-hyperemic pressure ratio (NHPR) metrics which allow rapid invasive coronary physiology measurements within seconds without the cost and potential side effects of adenosine administration associated with traditional hyperemic physiology measures, now offers the capability to routinely perform physiology guided PCI approach for visually severe lesions.

REFINE-PCI is a prospective, single-center study in which participants with coronary artery stenosis deemed severe by visual angiography and planned for PCI without physiology assessment will undergo blinded invasive physiologic measurements using a coronary-pressure sensing wire pre and post PCI (OpSens OptoWire III) to assess the physiologic significance of the stenosis. Participants will also complete a health-related quality of life survey pre and 30 days post stent placement to assess for clinical change following PCI.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Patient provides written informed consent
* Clinical presentation with stable coronary artery disease or acute coronary syndromes (unstable angina, Non-ST Elevation Myocardial Infarction (NSTEMI), or ST Elevation Myocardial Infarction (STEMI))
* Scheduled for clinically indicated cardiac catheterization
* At least one lesion with angiographic severity visually estimated to be >/= 70% diameter stenosis that is deemed suitable for PCI
* The operator plans to perform PCI on an ad hoc or planned basis
* The target lesion is not planned for assessment by invasive physiology

Exclusion Criteria:

* Failure to provide signed informed consent
* Culprit vessel of acute ST Elevation Myocardial Infarction (STEMI)
* Culprit vessel of Non-ST Elevation Myocardial Infarction (NSTEMI)
* Thrombolysis In Myocardial Infarction (TIMI) flow less than grade 3 at baseline or visible thrombus
* Chronic total occlusion (CTO) in the target vessel
* Target vessel is supplied by major collaterals or supplies major collaterals to a CTO
* Target lesion involves the left main coronary artery
* Prior history of coronary artery bypass grafting (CABG) to the target vessel, except if bypass graft is occluded
* Previously known untreated severe valvular heart disease
* Previously known left ventricular ejection fraction <30%
* Sustained ventricular arrhythmias
* Patients who are currently pregnant (pregnancy testing will be performed as per standard cardiac catheterization laboratory protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of male and female subjects from the general interventional cardiology population who are scheduled for coronary angiogram at Beth Israel Deaconess Medical Center
Sampling Method: Probability Sample
Enrollment: 107 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The percentage of physiologically non-significant lesions observed | Time of procedure
  Non-significant lesions defined as a diastolic pressure ratio (dPR) </= 0.89 (range 0-1), expressed as mean, standard deviation, and percentage of total number of assessments
Correlation of the operator visual angiographic assessment of stenosis severity with quantitative coronary angiography (QCA) and resting non-hyperemic pressure resting indices (NHPR) | Within 30 days post procedure
  Visual stenosis severity and QCA are numerical variables reported as percentages, and expressed as mean and standard deviation. NHPR is a numerical variable from 0 to 1, expressed as mean and standard deviation. Pearson correlation coefficient used to express correlation between two variables.
Correlation between QCA and NHPR | Within 30 days post procedure
  QCA is a numerical variable reported as a percentage, and expressed as mean and standard deviation. NHPR is a numerical variable from 0 to 1, expressed as mean and standard deviation. Pearson correlation coefficient used to express correlation between two variables.

SECONDARY OUTCOMES:
Correlation of the post-PCI NHPR with burden of angina as assessed via the Seattle Angina Questionnaire at 30 days post PCI | Day 30 post PCI
  NHPR is a numerical variable from 0 to 1, expressed as mean and standard deviation. Seattle Angina Questionnaire assesses patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, expressed as mean and standard deviation. Pearson correlation coefficient used to express correlation between two variables.
Change in angina as assessed via the Seattle Angina Questionnaire at baseline and 30 days after PCI, need for titration for anti-anginal medications, or need for repeat coronary angiography within 30 days of the procedure. | Day 30 post PCI
  Seattle Angina Questionnaire assesses patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life. Each scale is transformed to a score of 0 to 100, expressed as mean and standard deviation. Comparison of baseline and 30 days post PCI involves comparison of numerical variables and uses the Student's paired t test or Wilcoxon signed rank test. Need for titration for anti-anginal medications and need for repeat coronary angiography within 30 days of the procedure are descriptive data (Yes, No)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Osborn, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data collected is specific to this clinical trial question

REFERENCES:
- [Background] Davies JE, Sen S, Dehbi HM, Al-Lamee R, Petraco R, Nijjer SS, Bhindi R, Lehman SJ, Walters D, Sapontis J, Janssens L, Vrints CJ, Khashaba A, Laine M, Van Belle E, Krackhardt F, Bojara W, Going O, Harle T, Indolfi C, Niccoli G, Ribichini F, Tanaka N, Yokoi H, Takashima H, Kikuta Y, Erglis A, Vinhas H, Canas Silva P, Baptista SB, Alghamdi A, Hellig F, Koo BK, Nam CW, Shin ES, Doh JH, Brugaletta S, Alegria-Barrero E, Meuwissen M, Piek JJ, van Royen N, Sezer M, Di Mario C, Gerber RT, Malik IS, Sharp ASP, Talwar S, Tang K, Samady H, Altman J, Seto AH, Singh J, Jeremias A, Matsuo H, Kharbanda RK, Patel MR, Serruys P, Escaned J. Use of the Instantaneous Wave-free Ratio or Fractional Flow Reserve in PCI. N Engl J Med. 2017 May 11;376(19):1824-1834. doi: 10.1056/NEJMoa1700445. Epub 2017 Mar 18. PMID 28317458
- [Background] Gotberg M, Christiansen EH, Gudmundsdottir IJ, Sandhall L, Danielewicz M, Jakobsen L, Olsson SE, Ohagen P, Olsson H, Omerovic E, Calais F, Lindroos P, Maeng M, Todt T, Venetsanos D, James SK, Karegren A, Nilsson M, Carlsson J, Hauer D, Jensen J, Karlsson AC, Panayi G, Erlinge D, Frobert O; iFR-SWEDEHEART Investigators. Instantaneous Wave-free Ratio versus Fractional Flow Reserve to Guide PCI. N Engl J Med. 2017 May 11;376(19):1813-1823. doi: 10.1056/NEJMoa1616540. Epub 2017 Mar 18. PMID 28317438
- [Background] De Bruyne B, Pijls NH, Kalesan B, Barbato E, Tonino PA, Piroth Z, Jagic N, Mobius-Winkler S, Rioufol G, Witt N, Kala P, MacCarthy P, Engstrom T, Oldroyd KG, Mavromatis K, Manoharan G, Verlee P, Frobert O, Curzen N, Johnson JB, Juni P, Fearon WF; FAME 2 Trial Investigators. Fractional flow reserve-guided PCI versus medical therapy in stable coronary disease. N Engl J Med. 2012 Sep 13;367(11):991-1001. doi: 10.1056/NEJMoa1205361. Epub 2012 Aug 27. PMID 22924638
- [Background] Jeremias A, Davies JE, Maehara A, Matsumura M, Schneider J, Tang K, Talwar S, Marques K, Shammas NW, Gruberg L, Seto A, Samady H, Sharp A, Ali ZA, Mintz G, Patel M, Stone GW. Blinded Physiological Assessment of Residual Ischemia After Successful Angiographic Percutaneous Coronary Intervention: The DEFINE PCI Study. JACC Cardiovasc Interv. 2019 Oct 28;12(20):1991-2001. doi: 10.1016/j.jcin.2019.05.054. PMID 31648761
- [Background] Collison D, McClure JD, Berry C, Oldroyd KG. A randomized controlled trial of a physiology-guided percutaneous coronary intervention optimization strategy: Rationale and design of the TARGET FFR study. Clin Cardiol. 2020 May;43(5):414-422. doi: 10.1002/clc.23342. Epub 2020 Feb 10. PMID 32037592